CLINICAL TRIAL: NCT00610155
Title: A Methodology Study To Assess The Feasibility Of Using Functional Magnetic Resonance Imaging (fRMI) To Quantify The Effects Of Analgesic Drugs In Post-Traumatic Neuropathic Pain Subjects
Brief Title: A Methodology Study Of Brain Imaging Of Pain-Killers In Post-Traumatic Neuropathic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081173
Record Dates: First submitted 2008-01-14; First posted 2008-02-07 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2013-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Pregabalin
- 3 (Experimental)
  Interventions: Drug: Tramadol SR

INTERVENTIONS:
Drug: Placebo — BID
  Arms: 1
Drug: Pregabalin — Dose 75 mg titrated to 150 mg, bid
  Arms: 2
Drug: Tramadol SR — Dose 50mg titrated to 200 mg, bid
  Arms: 3

SUMMARY:
This study is a methodology study designed to discover whether a brain imaging technology is a better way of compare the relative sensitivities of fMRI and subjective psychometric assessments of pain to multiple doses of pregabalin and tramadol SR in a cross-over clinical study design.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neuropathic pain associated with brush allodynia in specific dermatomes.
* Brush allodynia score of ≥4 and calculated average pain score of ≥3 on an 11-point numerical rating scale by the completion of down-titration of existing medications.
* Right-handed

Exclusion Criteria:

* Subjects with trigeminal neuralgia, central pain (due to cerebrovascular lesions, multiple sclerosis and/or traumatic spinal cord injuries including spinal surgery).
* Phantom limb pain, painful diabetic neuropathy.
* Subjects with any other co-existing pain which he/she or a qualified pain physician cannot differentiate from NeP of peripheral origin.
* Subjects with diabetes mellitus and with an HbA1C value of >10% upon measurement at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United Kingdom (2):
  - Pfizer Investigational Site, Portsmouth, Hampshire
  - Pfizer Investigational Site, Solihull, West Midlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin Then Tramadol Then Placebo: Pregabalin (PGB) capsule titrated to 150 milligram (mg) orally twice daily for 7 days in first intervention period; followed by tramadol (TMD) sustained release (SR) capsule titrated to 200 mg orally twice daily for 7 days in second intervention period; then matching placebo (PBO) capsule orally for 7 days in third intervention period. A placebo wash-out period of 7 days was maintained between each period.
- Tramadol Then Placebo Then Pregabalin: Tramadol SR capsule titrated to 200 mg orally twice daily for 7 days in first intervention period; followed by matching placebo capsule orally for 7 days in second intervention period; then pregabalin capsule titrated to 150 mg orally twice daily for 7 days in third intervention period. A placebo wash-out period of 7 days was maintained between each period.
- Placebo Then Pregabalin Then Tramadol: Matching placebo capsule orally for 7 days in first intervention period; followed by pregabalin capsule titrated to 150 mg orally twice daily for 7 days in second intervention period; then tramadol SR capsule titrated to 200 mg orally twice daily for 7 days in third intervention period. A placebo wash-out period of 7 days was maintained between each period.
- Pregabalin Then Placebo Then Tramadol: Pregabalin capsule titrated to 150 mg orally twice daily for 7 days in first intervention period; followed by matching placebo capsule orally for 7 days in second intervention period; then tramadol SR capsule titrated to 200 mg orally twice daily for 7 days in third intervention period. A placebo wash-out period of 7 days was maintained between each period.
- Placebo Then Tramadol Then Pregabalin: Matching placebo capsule orally for 7 days in first intervention period; followed by tramadol SR capsule titrated to 200 mg orally twice daily for 7 days in second intervention period; then pregabalin capsule titrated to 150 mg orally twice daily for 7 days in third intervention period. A placebo wash-out period of 7 days was maintained between each period.
- Tramadol Then Pregabalin Then Placebo: Tramadol SR capsule titrated to 200 mg orally twice daily for 7 days in first intervention period; followed by pregabalin capsule titrated to 150 mg orally twice daily for 7 days in second intervention period; then matching placebo capsule orally for 7 days in third intervention period. A placebo wash-out period of 7 days was maintained between each period.
Period: Period 1
Arm/Group | Pregabalin Then Tramadol Then Placebo | Tramadol Then Placebo Then Pregabalin | Placebo Then Pregabalin Then Tramadol | Pregabalin Then Placebo Then Tramadol | Placebo Then Tramadol Then Pregabalin | Tramadol Then Pregabalin Then Placebo
Started | 4 | 3 | 4 | 3 | 3 | 1
Completed | 4 | 3 | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | Pregabalin Then Tramadol Then Placebo | Tramadol Then Placebo Then Pregabalin | Placebo Then Pregabalin Then Tramadol | Pregabalin Then Placebo Then Tramadol | Placebo Then Tramadol Then Pregabalin | Tramadol Then Pregabalin Then Placebo
Started | 4 | 3 | 3 | 3 | 3 | 1
Completed | 4 | 3 | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Pregabalin Then Tramadol Then Placebo | Tramadol Then Placebo Then Pregabalin | Placebo Then Pregabalin Then Tramadol | Pregabalin Then Placebo Then Tramadol | Placebo Then Tramadol Then Pregabalin | Tramadol Then Pregabalin Then Placebo
Started | 4 | 3 | 3 | 3 | 3 | 1
Completed | 4 | 3 | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | Pregabalin Then Tramadol Then Placebo | Tramadol Then Placebo Then Pregabalin | Placebo Then Pregabalin Then Tramadol | Pregabalin Then Placebo Then Tramadol | Placebo Then Tramadol Then Pregabalin | Tramadol Then Pregabalin Then Placebo
Started | 4 | 3 | 3 | 3 | 3 | 1
Completed | 4 | 3 | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Pregabalin Then Tramadol Then Placebo | Tramadol Then Placebo Then Pregabalin | Placebo Then Pregabalin Then Tramadol | Pregabalin Then Placebo Then Tramadol | Placebo Then Tramadol Then Pregabalin | Tramadol Then Pregabalin Then Placebo
Started | 4 | 3 | 3 | 3 | 3 | 1
Completed | 3 | 3 | 3 | 3 | 3 | 1
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants enrolled in the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Voxel-wise Blood Oxygen Level Dependent (BOLD) Using Functional Magnetic Resonance Imaging (fMRI) of Brain Activation Signals Across the Whole Brain
Description: BOLD brain activation signals in whole brain was assessed using Contrast Parameter Estimates (COPE) images in response to dynamic mechanical allodynia of the affected side (DMAa), dynamic mechanical allodynia of the control side (DMAc), thermal pain (TH) and checkerboard visual stimuli (VIS).
Time Frame: Day 8, 22, 36
Population: Data not available to report, as BOLD brain activation signals in whole brain were obtained as specific Contrast Parameter Estimates (COPE) images only, as per planned analysis.
Groups:
- Pregabalin: Pregabalin capsule titrated to 150 mg orally twice daily for 7 days in either of the intervention periods.
- Tramadol: Tramadol SR capsule titrated to 200 mg orally twice daily for 7 days in either of the intervention periods.
- Placebo: Matching placebo capsule orally for 7 days in either of the intervention periods.
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Voxel-wise Blood Oxygen Level Dependent (BOLD) Using fMRI of Brain Activation Signals in Defined Brain Regions in Response to Dynamic Mechanical Allodynia of the Affected Side (DMAa)
Description: BOLD brain activation signals in pre-defined region of interest(ROI):anterior cingulate cortex(ACC);left,right anterior cortex([AIC_L ],[AIC_R]);left,right mid-insular cortex([MIC_L],[MIC_R]);left,right posterior insular cortex([PIC_L],[PIC_R]);left,right amygdala([Amyg_L],[Amyg_R]);primary,secondary somatosensory cortex([S1],[S2]);sensory part of thalamus(SensTHAL);midbrain reticular formation(MRF);nucleus cuneiformis(NucCun);periaqueductal gray(PAG). Prior to ROI analysis, a prelimanary anlysis was performed, wherein it was concluded that ROI analysis was to be carried out for DMAa, DMAc amd TH only. In voxel BOLD analysis,signal change is unit less measure but approximated to percent signal change by grand scaling(effects divided by 10000 to get percent signal change).
Time Frame: Day 8, 22, 36
Population: BOLD analysis set included all participants who completed all the 3 treatment periods of the study.
Measure: Least Squares Mean (Standard Error); unit: percent signal change
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 16 | 16 | 16
percent signal change
  ACC | -17.3 (9.7) | 18.6 (9.7) | 7.4 (9.7)
  AIC_L | 8.1 (8.8) | 23.3 (8.8) | 30.8 (8.8)
  AIC_R | 11.1 (10.0) | 21.9 (10.0) | 17.1 (10.0)
  MIC_L | 3.8 (8.4) | 23.4 (8.4) | 30.0 (8.4)
  MIC_R | 8.6 (8.4) | 13.4 (8.4) | 18.3 (8.4)
  PIC_L | -6.8 (5.2) | -5.8 (5.2) | -0.3 (5.2)
  PIC_R | -13.6 (8.5) | 2.9 (8.5) | 6.5 (8.5)
  Amyg_L | -5.7 (10.2) | 5.5 (10.2) | 8.5 (10.2)
  Amyg_R | -1.4 (8.5) | 20.3 (8.5) | 21.7 (8.5)
  S1 | -28.5 (20.5) | -4.1 (20.5) | -2.9 (20.5)
  S2 | 2.5 (10.8) | -3.2 (10.8) | 10.8 (10.8)
  SensTHAL | 8.0 (5.4) | 16.5 (5.4) | 9.6 (5.4)
  MRF | 7.0 (5.0) | 6.4 (5.0) | 11.7 (5.0)
  NucCun | 1.1 (5.5) | -0.9 (5.5) | 12.9 (5.5)
  PAG | -3.8 (7.9) | -15.3 (7.9) | 2.5 (7.9)

3. Primary Outcome: Voxel-wise Blood Oxygen Level Dependent (BOLD) Using fMRI of Brain Activation Signals in Defined Brain Regions in Response to Dynamic Mechanical Allodynia of the Control Side (DMAc)
Description: BOLD brain activation signals in pre-defined ROI. ROI were ACC; AIC_L; AIC_R; MIC_L; MIC_R; PIC_L; PIC_R; Amyg_L; Amyg_R; S1; S2; SensTHAL; MRF; NucCun; PAG. Prior to ROI analysis, a prelimanary anlysis was performed, wherein it was concluded that ROI analysis was to be carried out for DMAa, DMAc amd TH only. In voxel BOLD analysis, signal change is unit less measure but is approximated to percent signal change here by grand scaling (dividing effects by 10000 to get percent signal change).
Time Frame: Day 8, 22, 36
Population: BOLD analysis set included all participants who completed all the 3 treatment periods of the study.
Measure: Least Squares Mean (Standard Error); unit: percent signal change
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 16 | 16 | 16
percent signal change
  ACC | -22.3 (12.0) | -3.7 (12.0) | 0.2 (12.0)
  AIC_L | -13.5 (8.0) | 18.2 (8.0) | 20.2 (8.0)
  AIC_R | -10.6 (7.4) | 10.3 (7.4) | 20.2 (7.4)
  MIC_L | -7.6 (8.4) | 9.7 (8.4) | 9.0 (8.4)
  MIC_R | -9.2 (6.2) | 2.8 (6.2) | 0.7 (6.2)
  PIC_L | -14.9 (6.9) | -8.1 (6.9) | 0.8 (6.9)
  PIC_R | -17.2 (9.4) | 2.4 (9.4) | 6.3 (9.4)
  Amyg_L | -14.3 (7.3) | 1.5 (7.3) | -3.4 (7.3)
  Amyg_R | -10.3 (9.7) | 2.0 (9.7) | -3.8 (9.7)
  S1 | -31.6 (16.2) | -4.5 (16.2) | 14.6 (16.2)
  S2 | -0.4 (8.3) | 9.6 (8.3) | 13.5 (8.3)
  SensTHAL | 3.9 (5.3) | -2.8 (5.3) | 6.7 (5.3)
  MRF | 1.5 (4.6) | -6.6 (4.6) | -1.7 (4.6)
  NucCun | 1.0 (4.9) | -8.2 (4.9) | -1.8 (4.9)
  PAG | 1.6 (7.8) | -12.0 (7.8) | -5.0 (7.8)

4. Primary Outcome: Voxel-wise Blood Oxygen Level Dependent (BOLD) Using fMRI of Brain Activation Signals in Defined Brain Regions in Response to Thermal Stimulation (TH)
Description: as for outcome 3
Time Frame: Day 8, 22, 36
Population: BOLD analysis set included all participants who completed all the 3 treatment periods of the study.
Measure: Least Squares Mean (Standard Error); unit: percent signal change
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 16 | 16 | 16
percent signal change
  ACC | 102.2 (25.9) | 92.5 (25.8) | 83.3 (25.8)
  AIC_L | 92.1 (21.9) | 103.4 (21.8) | 118.7 (21.8)
  AIC_R | 121.7 (20.7) | 104.6 (20.6) | 104.0 (20.6)
  MIC_L | 93.4 (19.6) | 105.2 (19.5) | 100.4 (19.5)
  MIC_R | 106.6 (17.3) | 71.1 (17.3) | 92.0 (17.3)
  PIC_L | 31.2 (16.0) | 44.6 (15.9) | 34.2 (15.9)
  PIC_R | 75.3 (20.1) | 95.5 (20.0) | 91.8 (20.0)
  Amyg_L | 29.7 (16.5) | 24.9 (16.5) | 36.4 (16.5)
  Amyg_R | 77.5 (22.5) | 57.2 (22.5) | 67.0 (22.5)
  S1 | -49.0 (30.2) | 37.7 (30.1) | 27.7 (30.1)
  S2 | 73.6 (21.2) | 94.6 (21.2) | 74.5 (21.2)
  SensTHAL | 19.4 (12.1) | 0.8 (12.1) | 10.4 (12.1)
  MRF | 34.3 (14.7) | 25.5 (14.6) | 37.7 (14.6)
  NucCun | 38.7 (11.5) | 27.7 (11.5) | 40.5 (11.5)
  PAG | 63.3 (15.9) | 53.6 (15.8) | 44.6 (15.8)

5. Primary Outcome: Voxel-wise Blood Oxygen Level Dependent (BOLD) Using fMRI of Brain Activation Signals in Defined Brain Regions in Response to Visual Stimulation (VIS)
Description: BOLD brain activation signals in pre-defined ROI in response to checkerboard visual stimuli (flashing at 2 Hz). ROI were ACC; AIC_L; AIC_R; MIC_L; MIC_R; PIC_L; PIC_R; Amyg_L; Amyg_R; S1; S2; SensTHAL; MRF; NucCun; PAG. Prior to ROI analysis, a prelimanary anlysis was performed, wherein it was concluded that ROI analysis was to be carried out for DMAa, DMAc amd TH only.
Time Frame: Day 8, 22, 36
Population: For VIS, based on preliminary analysis results, it was not considered significant to collect data according to Investigator's opinion.
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: Arterial Spin Labelling (ASL) Using fMRI of Brain Activation Signals Across the Whole Brain and in Defined Brain Regions
Description: Continuous ASL sequence fMRI imaging modality assessing brain activation signals across the whole brain and in defined ROI to assess effects of evoked pain along with changes in regional cerebral blood flow (rCBF). ROI were ACC; AIC_L; AIC_R; MIC_L; MIC_R; PIC_L; PIC_R; Amyg_L; Amyg_R; S1; S2; SensTHAL; MRF; NucCun; PAG.
Time Frame: Day 8, 22, 36
Population: Data was not analyzed since these methods were not technically robust enough to make any clear conclusions.
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36)
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Day 8, 22, 36
Population: Data for this outcome measure was plotted against treatment for each participant as per planned analysis but not statistically summarized for analysis.
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Beck Depression Inventory (BDI)
Description: BDI is a 21 item participant rated inventory evaluating depression symptoms, cognition, and physical symptoms of fatigue, weight loss, lack of interest in sex. Individual items are scored on a 4 point scale (0 to 3), with 0=none/absent and 3=most severe. Total score: 0 to 63; higher score indicate more depression.
Time Frame: Day 8, 22, 36
Population: as for outcome 7
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: State and Trait Anxiety Questionnaire
Description: Self-report scale completed by the participant. Separate scales measure state (20 items) and trait (20 items) anxiety. The participant report how they feel "right now at this moment" for state anxiety and how they "generally" feel for trait anxiety. The "state" items are scored as: 1 (not at all), 2 (somewhat true), 3 (moderately true), 4 (very much so). The "trait" items are scored as: 1 (almost never), 2 (sometimes), 3 (often), 4 (almost always). Scores range from 20-80 for each scale. Higher scores indicate more impaired participants.
Time Frame: Day 8, 22, 36
Population: as for outcome 7
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Pain Catastrophising Scale (PCS)
Description: The PCS is a self-administered questionnaire with 13 items, each scored from 0 (not at all) to 4 (all the time) for extent to which participant catastrophizes postoperative pain. Total score is sum of scores for all questions (range: 0 to 52); Subscale scores: Rumination (sum of scores for 4 items; range: 0 to 16); Magnification (sum of scores for 3 items; range: 0 to 12); and Helplessness (sum of scores for 6 items; range: 0 to 24); higher scores indicate greater extent of pain catastrophizing.
Time Frame: Day 8, 22, 36
Population: as for outcome 7
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Neuropathic Pain Symptom Inventory (NPSI)
Description: NPSI: participant rated questionnaire to evaluate different symptoms of neuropathic pain (dimensions: burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia [P/D]). Includes 10 descriptors quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. Questionnaire generates a score in each of the relevant dimensions and a total score of 0-100. Higher score indicate a greater intensity of pain.
Time Frame: Baseline (Day -7), Day 8, 22, 36
Population: as for outcome 7
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Daily Pain Score
Description: Daily Pain Score: Day 1 pain intensity over past 24 hours recorded on waking every morning using 0-10 numeric rating scale (NRS): 0 (no pain) to 10 (worst possible pain). The daily pain scores for an average of the last 7 days and an average of last 3 days were calculated.
Time Frame: Day -35 through Day 36
Population: FAS included all the participants who were enrolled in the study. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 18 | 17 | 18
units on a scale
  Last 7 days | 5.57 (0.371) | 5.28 (0.370) | 6.40 (0.370)
  Last 3 days | 5.46 (0.466) | 5.10 (0.454) | 6.33 (0.454)

13. Secondary Outcome: Present Pain Intensity Score (PPIS)
Description: Participants answered: "Please rate your pain from 0-10 that best describes the intensity of pain right now". PPIS assessed on 0-10 numeric rating scale (NRS), 0 (no pain) to 10 (worst possible pain).
Time Frame: Day 8, 22, 36
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 17 | 17 | 17
units on a scale | 5.54 (0.552) | 4.13 (0.551) | 5.83 (0.551)

14. Secondary Outcome: Doleur Neuropathic 4 (DN4) Score
Description: DN4 questionnaire provides a simple diagnosis of Neuropathic pain (NeP) by asking for yes/no answers to 4 questions (10 sub questions in total). Each question was scored on a scale of 0 (No) and 1 (Yes). Total score was calculated as sum of the 10 individual questions. Total score range 0-10, higher score indicated more neuropathic pain.
Time Frame: Day -35
Population: as for outcome 7
Arm/Group | Pregabalin | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. But, distinct events are presented. An event may be categorized as serious in 1 subject; as nonserious in another subject or 1 subject may have experienced both serious, nonserious events in study.'At risk population'=who received study treatments in different interventions;PGB=17,TMD=17,PBO=18.
Arm/Group | Pregabalin | Tramadol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 14/17 | 14/17 | 11/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=17) | Tramadol (N=17) | Placebo (N=18)
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 8 | 1
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 6 | 1
Feeling hot (General disorders) | 0 | 1 | 0
Feeling of body temperature change (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 1 | 1
Clumsiness (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 7 | 8 | 2
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 2 | 4 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Libido decreased (Psychiatric disorders) | 1 | 0 | 1
Loss of libido (Psychiatric disorders) | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Results for primary outcome, BOLD activation signals(whole brain) was not available to reported, as DMAa, DMAc, TH and VIS were captured as COPE images only, which could not be included in basic results format.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.